CLINICAL TRIAL: NCT01658124
Title: Tranexamic Acid for the Treatment of Gastrointestinal Haemorrhage: an International Randomised, Double Blind Placebo Controlled Trial
Brief Title: Haemorrhage Alleviation With Tranexamic Acid- Intestinal System
Acronym: HALT-IT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Rawalpindi Medical College (Other); University of Ibadan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ISRCTN11225767
Record Dates: First submitted 2012-07-26; First posted 2012-08-06 (Estimated); Last update posted 2020-04-17 (Actual); Status verified 2020-02

CONDITIONS: Gastrointestinal Bleeding
Keywords: haemorrhage,antifibrinolytic, clinical trial,
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tranexamic acid (Experimental): (total dose 8 grams)
  Interventions: Drug: Tranexamic Acid
- Placebo (Placebo Comparator): (Sodium Chloride 0.9%)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid
  Arms: Tranexamic acid
Drug: Placebo
  Arms: Placebo

SUMMARY:
Severe bleeding in the digestive system is a common symptom of many diseases. Each year, about 50,000 people end up in British hospitals because of this problem and about 5,000 of them die. The most common cause of this bleeding is stomach ulcers. In sub-Saharan Africa, schistosomiasis (parasitic worms) is responsible for about 130,000 deaths from stomach bleeding each year. From previous research in other bleeding conditions such as surgery and trauma, we know that a drug called tranexamic acid can reduce bleeding and save lives. We now want to do the HALT-IT trial to see if giving tranexamic acid can save lives and if there are any complications in people with severe bleeding from the digestive system.

DETAILED DESCRIPTION:
BACKGROUND: Acute gastrointestinal (GI) haemorrhage is one of the most common gastrointestinal emergencies. It is an important cause of mortality and morbidity in high, middle and low income countries. The most common causes of upper GI haemorrhage are peptic ulcer, oesophageal varices and erosive mucosal disease, although the relative frequency of the different causes varies in different countries. Acute upper GI haemorrhage accounts for around 50,000 hospital admissions each year in the UK and has a case fatality of about 10%. The incidence is highest among the most disadvantaged social groups. Lower GI haemorrhage accounts for a further 15,000 hospital admissions each year and has a case fatality of between 10% and 20%. Upper GI haemorrhage is also a common medical emergency in low and middle income countries. Patients are usually young and poor and the source of bleeding is more often oesophageal varices. Fibrinolysis may play an important pathological role in GI haemorrhage due to premature breakdown of haemostatic plugs at sites of mucosal injury. Tranexamic acid (TXA) is a synthetic derivative of the amino acid lysine which inhibits fibrinolysis by blocking the lysine binding sites on plasminogen. It is a widely used treatment with a known safety profile. There is reliable evidence that TXA reduces blood transfusion in surgical patients. A systematic review including 65 trials shows that TXA reduces the probability of blood transfusion by 39% (RR=0.61, 95% CI 0.53 to 0.70) compared to control. The effect of TXA on the risk of thromboembolic events in surgical patients remains uncertain, although there is no evidence of any increase in risk. The CRASH-2 trial showed that administration of TXA significantly reduces deaths due to bleeding (RR=0.85, 95% CI 0.76 to 0.96), and all-cause mortality (RR=0.91, 95% CI 0.85 to 0.97) in trauma patients with significant extra-cranial bleeding, with no increase in vascular occlusive events. A systematic review conducted by the investigators of TXA in GI bleeding identified nine randomised trials including a total of 1721 patients. Although there was a statistically significant reduction in the risk of death in patients treated with TXA (RR=0.66, 95% CI 0.47 to 0.93), the estimate is imprecise and the overall quality of trials was poor. Furthermore, all but three of the trials were conducted before the widespread use of therapeutic endoscopy and proton pump inhibitors and even in aggregate the trials were too small to assess the effects of TXA on other clinical important outcomes such as thromboembolic events. For these reasons, the effectiveness and safety of TXA for GI haemorrhage is uncertain and there are currently no formal recommendations for its use as a treatment for GI bleeding.

AIM: The HALT-IT trial will determine the effect of TXA on mortality, morbidity (re-bleeding, non-fatal vascular events), blood transfusion, surgical intervention and health status in patients with acute gastrointestinal haemorrhage.

PRIMARY OUTCOME: The primary outcome is death from haemorrhage within 5 days of randomisation (all cause and cause-specific mortality will also be recorded).

SECONDARY OUTCOMES:

1. Re-bleeding
2. Endoscopic, radiological or surgical intervention
3. Blood transfusion - blood or blood component units transfused
4. Thromboembolic events (myocardial infarction, stroke, pulmonary embolism, deep vein thrombosis)
5. Other adverse medical events (including renal failure, significant cardiac event, respiratory failure, hepatic failure, sepsis, pneumonia, seizure and other reported events)
6. Functional status measured using the Katz Index of Independence in Activities of Daily Living
7. Time spent at an intensive care unit
8. Length of stay in hospital
9. Patient status (death, hospital readmission) at 12 months will be ascertained if appropriate databases are available in the recruiting country

TRIAL DESIGN:

A pragmatic, randomised, double blind, placebo controlled trial among 12,000 patients with clinically significant gastrointestinal bleeding

DIAGNOSIS AND INCLUSION/EXCLUSION CRITERIA:

Adults with acute significant upper or lower gastrointestinal bleeding. The diagnosis of significant bleeding is clinical but may include patients with hypotension, tachycardia, or those likely to need transfusion, urgent endoscopy or surgery. The fundamental eligibility criterion is the responsible clinician's 'uncertainty' as to whether or not to use tranexamic acid in a particular patient with gastrointestinal bleeding. If the clinician believes there is a clear indication for, or clear contraindication to, tranexamic acid use, the particular patient should not be randomised. There are no other pre-specified exclusion criteria.

TEST PRODUCT, REFERENCE THERAPY, DOSE AND MODE OF ADMINISTRATION:

A loading dose of tranexamic acid (1 gram by intravenous injection) or placebo (sodium chloride 0.9%) will be given as soon as possible after randomisation followed by an intravenous infusion of 3 grams over 24 hours or placebo (sodium chloride 0.9%).

SETTING:

This trial will be coordinated from the London School of Hygiene & Tropical Medicine Clinical Trials Unit (University of London) and conducted in hospitals in low, middle and high income countries.

DURATION OF TREATMENT AND PARTICIPATION:

The first dose will be given immediately after randomisation and the maintenance dose will be given immediately after the loading dose over 24 hours. Participation will end at discharge from randomising hospital, death or at 28 days post randomisation whichever occurs first.

CRITERIA FOR EVALUATION:

All patients randomly assigned to one of the treatments will be analysed together (regardless of whether or not they completed or received that treatment) on an intention to treat basis.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* with acute significant upper or lower gastrointestinal bleeding
* where the responsible clinician is substantially uncertain as to the appropriateness of antifibrinolytic agents in the patient

Exclusion Criteria:

* The fundamental eligibility criterion is the responsible clinician's 'uncertainty' as to whether or not to use an antifibrinolytic agent in a particular patient with upper or lower gastrointestinal bleeding.
* There are no other exclusions.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12009 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2019-07-19 (Actual); Study Completion 2019-07-19 (Actual)

PRIMARY OUTCOMES:
The primary outcome is death from haemorrhage | within 5 days of randomisation

SECONDARY OUTCOMES:
Death (all cause and cause specific) | within 28 days of randomisation
Death from haemorrhage | within 28 days of randomisation
Number of Patients with Re-bleeding | within 5 and 28 days of randomisation
Number of patients who had Endoscopic, radiological or surgical intervention for gastro intestinal bleeding | within 28 days of randomisation
Number of patients who had Blood transfusion | within 28 days of randomisation
  blood or blood component units
Number of patients with Thromboembolic events | within 28 days of randomisation
  fatal and non-fatal myocardial infarction, stroke, pulmonary embolism, deep vein thrombosis
Number of patients with Other adverse medical events | within 28 days of randomisation
  including renal failure, significant cardiac event, respiratory failure, hepatic failure, sepsis, pneumonia, seizure, other reported events
Functional status measured using the Katz Index of Independence in Activities of Daily Living | within 28 days of randomisation
Time spent at an intensive care or high dependency unit | within 28 days of randomisation
Length of stay in hospital | within 28 days of randomisation
Patient status (death, hospital readmission) | within 12 months of randomisation
  Limited to recruiting countries with appropriate databases

CONTACTS AND LOCATIONS:
Overall Officials: Haleema Shakur-Still, Study Director — London School of Hygiene and Tropical Medicine
Locations (1):
- Over 50 countries Worldwide, London, United Kingdom

REFERENCES:
- [Derived] Roberts I, Shakur-Still H, Afolabi A, Akere A, Arribas M, Austin E, Bal K, Bazeer N, Beaumont D, Brenner A, Carrington L, Chaudhri R, Coats T, Gilmore I, Halligan K, Hussain I, Jairath V, Javaid K, Kayani A, Lisman T, Mansukhani R, Miners A, Mutti M, Nadeem MA, Pollok R, Prowse D, Simmons J, Stanworth S, Veitch A, Williams J. A high-dose 24-hour tranexamic acid infusion for the treatment of significant gastrointestinal bleeding: HALT-IT RCT. Health Technol Assess. 2021 Oct;25(58):1-86. doi: 10.3310/hta25580. PMID 34663491
- [Derived] HALT-IT Trial Collaborators. Effects of a high-dose 24-h infusion of tranexamic acid on death and thromboembolic events in patients with acute gastrointestinal bleeding (HALT-IT): an international randomised, double-blind, placebo-controlled trial. Lancet. 2020 Jun 20;395(10241):1927-1936. doi: 10.1016/S0140-6736(20)30848-5. PMID 32563378
- [Derived] Brenner A, Afolabi A, Ahmad SM, Arribas M, Chaudhri R, Coats T, Cuzick J, Gilmore I, Hawkey C, Jairath V, Javaid K, Kayani A, Mutti M, Nadeem MA, Shakur-Still H, Stanworth S, Veitch A, Roberts I; HALT-IT Trial Collaborators. Tranexamic acid for acute gastrointestinal bleeding (the HALT-IT trial): statistical analysis plan for an international, randomised, double-blind, placebo-controlled trial. Trials. 2019 Jul 30;20(1):467. doi: 10.1186/s13063-019-3561-7. PMID 31362765
- [Derived] Roberts I, Coats T, Edwards P, Gilmore I, Jairath V, Ker K, Manno D, Shakur H, Stanworth S, Veitch A. HALT-IT--tranexamic acid for the treatment of gastrointestinal bleeding: study protocol for a randomised controlled trial. Trials. 2014 Nov 19;15:450. doi: 10.1186/1745-6215-15-450. PMID 25409738
- See also: Trial website — http://haltit.lshtm.ac.uk/